CLINICAL TRIAL: NCT01506076
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Oral Dose, Crossover, Bioequivalence Study of Levocetirizine DiHCl Tablets 5mg With XYZAL® Tablets 5 mg in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Levocetirizine DiHCl Tablets 5mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07446/07-08
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levocetirizine DiHCl Tablets, 5 mg (Experimental): Levocetirizine DiHCl Tablets, 5 mg of Dr. Reddy's Laboratories Ltd.
  Interventions: Drug: Levocetirizine DiHCl
- XYZAL (Active Comparator): XYZAL Tablets 5 mg of UCB Farchim S.A.
  Interventions: Drug: Levocetirizine DiHCl

INTERVENTIONS:
Drug: Levocetirizine DiHCl — Levocetirizine DiHCl Tablets 5 mg
  Other Names: XYZAL

SUMMARY:
The purpose of this study is to assess the Bioequivalence of Levocetirizine DiHCl Tablets 5mg with XYZAL tablets 5 mg and to monitor clinical status, adverse events and laboratory investigations and assess relative safety and tolerance, under fasting conditions.

DETAILED DESCRIPTION:
A pivotal study to compare the Bioequivalence of Levocetirizine DiHCl Tablets 5 mg of Dr.Reddy's Laboratories Limited with XYZAL® Tablets 5 mg of UCB Farchim S.A. in healthy, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will provide written informed consent.
* Subjects must be healthy adults within 18-45 years of age (inclusive).
* Body mass index of ≥18.5 kg/m2 and ≤25 kg/m2, with body weight not less than 50 kg.
* Subjects must be of normal health as determined by medical history and physical examination performed within 15 days prior to the commencement of the dosing in Period-I.
* Have normal ECG, chest X-Ray and vital signs and clinically non significant changes in ECG & chest X-Ray.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
* Subjects will be Non smokers or moderate smokers (less than 10 cigarettes a day) for at least 6 months.
* If subject is a female volunteer and is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device(IUD), or abstinence.

or is postmenopausal for at least 1 year. is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

•Each female subject will be given a urine pregnancy test at screening, check-in for period-1, period-2 and post study.

Exclusion Criteria:

* Subjects incapable of understanding the informed consent.
* Subjects with BP lesser than 90/60 mm of Hg or BP greater than or equal to 140/90 mm of Hg.
* History of hypersensitivity or idiosyncratic reaction to Levocetirizine or other related drugs.
* Any evidence of impairment of renal, hepatic, gastro intestinal, lung and cardiac function.
* Subjects with a history of tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for the study.
* Regular smoker who smokes more than ten cigarettes daily or has difficulty in abstaining from smoking for the duration of each study period.
* Subjects who have taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication within the past two weeks prior to prior to dosing in Period-1.
* History of any psychiatric illness, which may impair the ability to provide written, informed consent.
* Subject is mentally or legally incapacitated, or has a history of significant psychiatric disorder.
* Subjects who have a history of alcohol or substance/ drug of abuse within the last 5 years.
* Subjects with clinically significant abnormal values of laboratory parameters, including positive results of HIV, HBV, HCV, RPR tests.
* Subjects who participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
* Subjects who are unable to or likely to be non-compliant with protocol requirements or restrictions.
* Subjects who are intolerant to venipuncture.
* Any subject in whom Levocetirizine Dihydrochloride is contraindicated for medical reasons.
* Female volunteers who has used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 14 days before dosing.
* Female volunteers demonstrating a positive pregnancy screen.
* All female subjects will be screened for pregnancy at screening, check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
* Female volunteers who are currently breast feeding. Female subjects who are pregnant, breast-feeding or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate.
* Subjects with positive urine screen for drugs of abuse at the time of admission check-in for each period will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Sudershan Vishwanath, MD, Principal Investigator — Vimta Labs Ltd.,
Locations (1):
- Vimta Labs Ltd.,, Hyderabad, A.P, India